CLINICAL TRIAL: NCT03632291
Title: A Phase I, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Dose of UB-221 as an Add-on Therapy in Patients With Chronic Spontaneous Urticaria
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of UB-221 as an Add-on Therapy in CSU Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A107-IgE
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Urticaria Chronic
Keywords: UB-221; anti-IgE monoclonal antibody; chronic spontaneous urticaria (CSU)
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- UB-221 (0.2 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (0.6 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (2 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (6 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221
- UB-221 (10 mg/kg) (Experimental): Intravenous infusion
  Interventions: Biological: UB-221

INTERVENTIONS:
Biological: UB-221 — UB-221 (75 mg/ml)

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single dose of UB-221 as an add-on therapy in patients with Chronic Spontaneous Urticaria.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single dose of UB-221 as an add-on therapy in patients with Chronic Spontaneous Urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age between 20 to 65 years old (inclusive).
* Subjects who are able and willing to provide the informed consent.
* Male subjects with body weight of 50 kilogram (kg) or above; female subjects body weight of 45 kilogram (kg) or above.
* Subjects diagnosed with chronic spontaneous urticaria (CSU).

Exclusion Criteria:

* History of significant diseases (other than CSU) or major clinical conditions by the investigator's judgment, such as auto-immune disease or psychiatric and behavioral conditions from which the investigator considers the subject is not suitable to participate in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | 15 days
  from the baseline to day 15 after IP infusion

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No